CLINICAL TRIAL: NCT00461305
Title: A Multicenter, Single-blind, Randomized Study, to Investigate Efficacy of Ethinylestradiol for Intracyclic Bleeding Profile During 24 Weeks (6 Cycles) by Oral Administration of Drospirenone 3 mg/Ethinylestradiol 20 µg and Drospirenone 3 mg/ Ethinylestradiol 30 µg in Patients With Dysmenorrheal and to Investigate the Long Term Safety Oral Administration of Drospirenone 3 mg/Ethinylestradiol 20 µg Administered for 52 Weeks (13 Cycles)
Brief Title: Safety Study of Ethinylestradiol/Drospirenone in Dysmenorrhea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Yakuhin, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91616; 310284 (Other: Company Internal)
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Intracyclic bleeding; Drospirenone (DRSP); Ethinylestradiol
MeSH Terms: conditions — Dysmenorrhea | interventions — drospirenone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRSP 3 mg/EE 20 µg (13 cycles) (Experimental): 1 tablet per day Drospirenone (DRSP) 3 mg/Ethinylestradiol (EE) 20 µg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle; treatment duration 52 weeks (13 cycles)
  Interventions: Drug: DRSP 3 mg/EE 20 µg (13 cycles)
- DRSP 3 mg/EE 30 µg (6 cycles) (Experimental): 1 tablet per day Drospirenone 3 mg/Ethinylestradiol 30 µg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle; treatment duration 24 weeks (6 cycles)
  Interventions: Drug: DRSP 3 mg/EE 30 µg (6 cycles)

INTERVENTIONS:
Drug: DRSP 3 mg/EE 20 µg (13 cycles) — 1 tablet per day Drospirenone (DRSP) 3 mg/Ethinylestradiol (EE) 20 µg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle; treatment duration 52 weeks (13 cycles)
  Arms: DRSP 3 mg/EE 20 µg (13 cycles)
Drug: DRSP 3 mg/EE 30 µg (6 cycles) — 1 tablet per day Drospirenone 3 mg/Ethinylestradiol 30 µg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle; treatment duration 24 weeks (6 cycles)
  Arms: DRSP 3 mg/EE 30 µg (6 cycles)

SUMMARY:
The purpose of this study is to investigate efficacy of ethinylestradiol for intracyclic bleeding profile in patients with dysmenorrhea and to investigate the long term safety

DETAILED DESCRIPTION:
The "drospirenone 3 mg/ethinylestradiol 20 μg (13 cycles)" group is to be treated by oral administration for 52 weeks, 13 cycles. The "drospirenone 3 mg/ethinylestradiol 30 μg (6 cycles)" group is to be treated by oral administration for 24 weeks, 6 cycles.

The trial is sponsored by Bayer Yakuhin, Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older at obtaining informed consent
* Patients having the normal menstrual cycle (25 to 38 days) in the latest two menses before the final enrollment
* Patients having a total dysmenorrheal score of at least 3 points in twice of the latest menstruation before the final enrollment

Exclusion Criteria:

* Patients with ovarian chocolate cysts
* Patients with fibroid needed to be treated
* Patients with estrogen-dependent tumors and patients with cervical cancer or suspected cervical cancer
* Patients with undiagnosed abnormal vaginal bleeding
* Patients with thrombophlebitis, pulmonary embolism, cerebrovascular disease, or coronary artery disease or a history of those diseases
* Patients aged 35 years or older who smoke at least 15 cigarettes per day
* Patients with migraine accompanied by prodromata
* Patients with pulmonary hypertension or valvular heart disease
* Patients who are regularly taking nutritional products that contain St. John's Wort
* Patients who underwent surgical treatment for endometriosis within 2 months prior to screening
* Patients who may need to regularly use analgesics for therapeutic objectives other than relief from the pain of dysmenorrhea during this study (occasional use permitted)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Japan (20):
  - Nagoya, Aichi-ken
  - Maebashi, Gunma
  - Takasaki, Gunma
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Yamato, Kanagawa
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Osaka, Osaka
  - Toyonaka, Osaka
  - Chuo-ku, Tokyo
  - Hachiōji, Tokyo
  - Machida, Tokyo
  - Musashino, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Suginami-ku, Tokyo
  - Toshima-ku, Tokyo

REFERENCES:
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS) consisted of all patients randomized who received at least one dose of study drug. Patients were analyzed as treated. FAS was the primary analysis set for the efficacy and safety. Per Protocol Set (PPS) was a subgroup of the FAS. The PPS consisted of patients in the FAS without major protocol deviations reported by Cycle 6.
Period: Treatment
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Started | 355 (Enrolled) | 65 (Enrolled)
Subjects Dispensed Drugs | 350 | 65
Subjects Received Treatment | 349 (FAS, safety population) | 65 (FAS, safety population)
Completed | 254 | 56
Not Completed | 101 | 9
Not completed — Adverse Event | 26 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 13 | 2
Not completed — Withdrawal by Subject | 48 | 2
Not completed — Never dispensed | 5 | 0
Not completed — Study drug not taken | 1 | 0
Not completed — Partially missing diary | 2 | 0
Not completed — Other (missing drug etc) | 2 | 0
Period: Continued Treatment
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Started | 349 (FAS, participants from previous treatment who were available to continue treatment) | 0 (no participants were treated with the DRSP 3 mg/EE 30 μg combination beyond 6 cycles)
Completed | 254 | 0
Not Completed | 95 | 0
Not completed — Adverse Event | 26 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Protocol Violation | 13 | 0
Not completed — Withdrawal by Subject | 48 | 0
Not completed — Partially missing diary | 2 | 0
Not completed — Other (missing drug etc) | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles) | Total
Number analyzed (Participants) | 349 | 65 | 414
Age Continuous [Mean (Full Range); unit: years] | 29.0 [20 to 44] | 30.9 [20 to 43] | 29.3 [20 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 65 | 414
  Male | 0 | 0 | 0
Diagnosis type [Number; unit: participants]
  Functional dysmenorrhea | 273 | 53 | 326
  Organic dysmenorrhea | 76 | 12 | 88
Details of organic dysmenorrhea [Number; unit: participants] — Not all participants had organic dysmenorrhea. Some of participants were diagnosed as having a multiple type of organic dysmenorrhea.
  participants
    Endometriosis | 24 | 4 | 28
    Uterine fibroids | 27 | 7 | 34
    Uterine adenomyosis | 35 | 8 | 43
    Endometrial polyp | 1 | 0 | 1
    Bicornuate uterus | 3 | 0 | 3
    Multiple endometrial polyp | 1 | 0 | 1
    Uterine enlargement | 1 | 0 | 1
Average length of menstrual cycle [Mean (Full Range); unit: days] | 29.5 [25 to 38] | 29.5 [25 to 38] | 29.5 [25 to 38]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 20.73 [16.2 to 29.9] | 20.56 [15.3 to 28.7] | 20.70 [15.3 to 29.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intracyclic Bleeding at Cycle 6
Description: Intracyclic bleedings were defined as bleedings while a participant takes active tablets.
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Groups:
- DRSP 3 mg/EE 20 µg (6 Cycles): 1 tablet per day Drospirenone (DRSP) 3 mg/Ethinylestradiol (EE) 20 µg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle; treatment duration 24 weeks (6 cycles)
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 299 | 56
participants | 40 | 4
Statistical Analysis 1: Comparison: DRSP 3 mg/EE 20 µg (6 Cycles); Exact 95% confident intervals were calculated using F-distribution by treatment group. If the upper confidence limit is lower than 27.56% (threshold incidence), the treatment arm will be concluded to be acceptable. No group comparison was planned; Test type: Superiority or Other; Binominal parameter by exact method; Incidence on one treatment arm = 13.4, 95% CI 2-sided [9.73 to 17.77] — No group comparison were planned. Binomial parameter on each treatment arm was estimated by exact method
Statistical Analysis 2: Comparison: DRSP 3 mg/EE 30 µg (6 Cycles); Exact 95% confident intervals were calculated using F-distribution by treatment group; Test type: Superiority or Other; Binominal parameter by exact method; Incidence on one treatment arm = 7.1, 95% CI [1.98 to 17.29]

2. Secondary Outcome: Number of Participants With a Change in Total Dysmenorrhea Score From Baseline to Cycle 6
Description: Total dysmenorrheal score was defined as sum of 2 sub-scores: severity of dysmenorrhea (none: 0, mild: 1, moderate: 2, severe: 3) and use of analgesics (none: 0, mild: 1, moderate: 2, severe: 3). Note: used with permission of Nobelpharma Co., Ltd. from the phase 3 clinical study protocol of IKH-01 in dysmenorrhea (associated with endometriosis) (Nobelpharma Co., Ltd.). Changed total dysmenorrheal scores: -6 to -1 mean improvement, 1 to 6 mean worsening, 0 means no change.
Time Frame: From baseline up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  -6 (change in total dysmenorrhea scores) | 5 | 2
  -5 (change in total dysmenorrhea scores) | 22 | 3
  -4 (change in total dysmenorrhea scores) | 41 | 8
  -3 (change in total dysmenorrhea scores) | 70 | 13
  -2 (change in total dysmenorrhea scores) | 71 | 10
  -1 (change in total dysmenorrhea scores) | 30 | 12
  0 (change in total dysmenorrhea scores) | 25 | 4
  1 (change in total dysmenorrhea scores) | 4 | 2
  2 (change in total dysmenorrhea scores) | 4 | 0
  3 (change in total dysmenorrhea scores) | 0 | 0
  4 (change in total dysmenorrhea scores) | 0 | 0
  5 (change in total dysmenorrhea scores) | 0 | 0
  6 (change in total dysmenorrhea scores) | 0 | 0

3. Secondary Outcome: Number of Participants With a Change in Total Dysmenorrhea Score From Baseline to Cycle 13
Description: as for outcome 2
Time Frame: From baseline up to Cycle 13 (364 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 13, note: no participants were treated with the DRSP 3 mg/EE 30 µg combination beyond 6 cycles)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  -6 (change in total dysmenorrhea scores) | 4
  -5 (change in total dysmenorrhea scores) | 22
  -4 (change in total dysmenorrhea scores) | 47
  -3 (change in total dysmenorrhea scores) | 68
  -2 (change in total dysmenorrhea scores) | 44
  -1 (change in total dysmenorrhea scores) | 32
  0 (change in total dysmenorrhea scores) | 12
  1 (change in total dysmenorrhea scores) | 11
  2 (change in total dysmenorrhea scores) | 2
  3 (change in total dysmenorrhea scores) | 0
  4 (change in total dysmenorrhea scores) | 0
  5 (change in total dysmenorrhea scores) | 0
  6 (change in total dysmenorrhea scores) | 0

4. Secondary Outcome: Distribution of Total Dysmenorrhea Score at Cycle 6
Description: Total dysmenorrhea score was defined as sum of 2 sub-scores: severity of dysmenorrhea and use of analgesics. Higher score means it is more severe. 0=None, 6=Severest.
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  0 | 65 | 13
  1 | 79 | 16
  2 | 49 | 9
  3 | 42 | 8
  4 | 19 | 3
  5 | 17 | 4
  6 | 1 | 1

5. Secondary Outcome: Distribution of Total Dysmenorrhea Score at Cycle 13
Description: as for outcome 4
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  0 | 73
  1 | 66
  2 | 41
  3 | 24
  4 | 24
  5 | 13
  6 | 1

6. Secondary Outcome: Distribution of Severity of Lower Abdominal Pain During Menstruation at Cycle 6
Description: Severity of lower abdominal pain during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  none | 75 | 14
  mild | 119 | 19
  moderate | 59 | 16
  severe | 19 | 5

7. Secondary Outcome: Distribution of Severity of Lower Abdominal Pain During Menstruation at Cycle 13
Description: as for outcome 6
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  none | 78
  mild | 106
  moderate | 47
  severe | 11

8. Secondary Outcome: Distribution of Severity of Lumbago During Menstruation at Cycle 6
Description: Severity of lumbago during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  none | 154 | 21
  mild | 88 | 29
  moderate | 26 | 2
  severe | 4 | 2

9. Secondary Outcome: Distribution of Severity of Lumbago During Menstruation at Cycle 13
Description: as for outcome 8
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  none | 148
  mild | 72
  moderate | 19
  severe | 3

10. Secondary Outcome: Distribution of Severity of Headache During Menstruation at Cycle 6
Description: Severity of headache during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  none | 187 | 37
  mild | 41 | 4
  moderate | 29 | 11
  severe | 15 | 2

11. Secondary Outcome: Distribution of Severity of Headache During Menstruation at Cycle 13
Description: as for outcome 10
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  none | 168
  mild | 38
  moderate | 30
  severe | 6

12. Secondary Outcome: Distribution of Severity of Nausea or Vomiting During Menstruation at Cycle 6
Description: Severity of nausea or vomiting during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
participants
  none | 251 | 51
  mild | 14 | 1
  moderate | 4 | 2
  severe | 3 | 0

13. Secondary Outcome: Distribution of Severity of Nausea or Vomiting During Menstruation at Cycle 13
Description: as for outcome 12
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  none | 229
  mild | 11
  moderate | 2
  severe | 0

14. Secondary Outcome: Number of Participants With a Total Pelvic Pain Score of 0 up to 6 at Times Other Than During Menstruation at Cycle 6
Description: Total pelvic pain score was defined as sum of 2 sub-scores: severity of dysmenorrhea and use of analgesics. Higher score means it is more severe. 0=None, 6=Severest.
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 271 | 54
participants
  0 | 202 | 34
  1 | 52 | 13
  2 | 11 | 4
  3 | 2 | 1
  4 | 2 | 1
  5 | 2 | 0
  6 | 0 | 1

15. Secondary Outcome: Number of Participants With a Total Pelvic Pain Score of 0 up to 6 at Times Other Than During Menstruation at Cycle 13
Description: as for outcome 14
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
participants
  0 | 177
  1 | 49
  2 | 12
  3 | 2
  4 | 2
  5 | 0
  6 | 0

16. Secondary Outcome: Change in Visual Analogue Scale (VAS) for Dysmenorrhea at Times Other Than During Menstruation From Baseline to Cycle 6
Description: VAS is an unmarked scale on a line 100 mm in length, indicating from 0 mm (no pain) to 100 mm (worst pain a participant has ever experienced).
Time Frame: From baseline up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 272 | 54
scores on a scale | -37.2 [-91 to 47] | -31.9 [-71 to 13]

17. Secondary Outcome: Change in Visual Analogue Scale (VAS) for Dysmenorrhea at Times Other Than During Menstruation From Baseline to Cycle 13
Description: as for outcome 16
Time Frame: From baseline up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
scores on a scale | -41.6 [-91 to 36]

18. Secondary Outcome: Change in Visual Analogue Scale (VAS) for Pelvic Pain at Times Other Than During Menstruation From Baseline to Cycle 6
Description: as for outcome 16
Time Frame: From baseline up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 271 | 54
scores on a scale | 6.7 [0 to 80] | 12.2 [0 to 83]

19. Secondary Outcome: Change in Visual Analogue Scale (VAS) for Pelvic Pain at Times Other Than During Menstruation From Baseline to Cycle 13
Description: as for outcome 16
Time Frame: From baseline up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 242
scores on a scale | 6.2 [0 to 65]

20. Secondary Outcome: Number of Any Bleeding Episodes From Cycle 1 to Cycle 6
Description: Vaginal bleeding was rated as none, spotting, light, normal, or heavy based on the participant's experience. A reference period is about 3 cycles (90 days): reference period 1 is from Cycle 1 to Cycle 3 (the 1st 90 days), reference period 2 is from Cycle 4 to Cycle 6 (the 2nd 90 days).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with the defined data, values for Cycle 1 to Cycle 6 (Reference period 1 and Reference period 2) in the DRSP 3mg/EE 20 µg group were calculated based on incomplete data due to the cut-off date)
Measure: Mean (Full Range); unit: number of episodes
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 326 | 60
number of episodes
  Reference period 1 | 3.3 [1 to 7] | 3.4 [1 to 7]
  Reference period 2 | 3.3 [0 to 10] | 3.1 [2 to 7]

21. Secondary Outcome: Number of Any Bleeding Episodes From Cycle 1 to Cycle 13
Description: Vaginal bleeding was rated as none, spotting, light, normal, or heavy based on the participant's experience. A reference period is about 3 cycles (90 days): reference period 1 is from Cycle 1 to Cycle 3 (the 1st 90 days), reference period 2 is from Cycle 4 to Cycle 6 (the 2nd 90 days), reference period 3 is from Cycle 7 to Cycle 9 (the 3rd 90 days), reference period 4 is from Cycle 10 to Cycle 12 (the 4th 90 days).
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: FAS (Participants with the defined data, note: no participants were treated with the DRSP 3 mg/EE 30 µg combination beyond 6 cycles)
Measure: Mean (Full Range); unit: number of episodes
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 333
number of episodes
  Reference period 1 | 3.2 [1 to 7]
  Reference period 2 | 3.5 [0 to 10]
  Reference period 3 | 3.1 [0 to 8]
  Reference period 4 | 3.2 [0 to 8]

22. Secondary Outcome: Number of Any Bleeding Days From Cycle 1 to Cycle 6
Description: as for outcome 20
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: as for outcome 20
Measure: Mean (Full Range); unit: days
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 326 | 60
days
  Reference period 1 | 30.7 [14 to 65] | 28.9 [13 to 65]
  Reference period 2 | 19.3 [0 to 78] | 19.9 [9 to 42]

23. Secondary Outcome: Number of Any Bleeding Days From Cycle 1 to Cycle 13
Description: Vaginal bleeding was rated as none, spotting, light, normal, or heavy based on the participant's experience. A reference period is about 3 cycles (90 days): reference period 1 is from Cycle 1 to Cycle 4 (the 1st 90 days), reference period 2 is from Cycle 4 to Cycle 6 (the 2nd 90 days), reference period 3 is from Cycle 7 to Cycle 9 (the 3rd 90 days), reference period 4 is from Cycle 10 to Cycle 12 (the 4th 90 days).
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 21
Measure: Mean (Full Range); unit: days
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 337
days
  Reference period 1 | 30.6 [14 to 65]
  Reference period 2 | 19.8 [0 to 79]
  Reference period 3 | 21.2 [0 to 88]
  Reference period 4 | 17.7 [0 to 69]

24. Secondary Outcome: Number of Participants With Intracyclic Bleeding From Cycle 1 to Cycle 6
Description: Intracyclic bleedings were defined as bleedings while a participant takes active tablets.
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS (Participants with data at Cycle 6, values for Cycle 1 to Cycle 6 (Reference period 1 and Reference period 2) in the DRSP 3mg/EE 20 µg group were calculated based on incomplete data due to the cut-off date)
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 341 | 62
participants
  Cycle 1 | 94 | 19
  Cycle 2 | 38 | 8
  Cycle 3 | 45 | 8
  Cycle 4 | 33 | 3
  Cycle 5 | 40 | 5
  Cycle 6 | 29 | 4

25. Secondary Outcome: Number of Participants With Intracyclic Bleeding From Cycle 1 to Cycle 13
Description: Intracyclic bleedings were defined as bleedings while a participant takes active tablets.
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 343
participants
  Cycle 1 | 93
  Cycle 2 | 38
  Cycle 3 | 45
  Cycle 4 | 33
  Cycle 5 | 41
  Cycle 6 | 40
  Cycle 7 | 114
  Cycle 8 | 24
  Cycle 9 | 24
  Cycle 10 | 24
  Cycle 11 | 21
  Cycle 12 | 23
  Cycle 13 | 31

26. Secondary Outcome: Number of Participants With Withdrawal Bleeding From Cycle 1 to Cycle 6
Description: Withdrawal bleedings were defined as bleedings while a participant takes placebo tablets.
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 341 | 62
participants
  Cycle 1 | 276 | 54
  Cycle 2 | 310 | 57
  Cycle 3 | 302 | 58
  Cycle 4 | 290 | 54
  Cycle 5 | 279 | 54
  Cycle 6 | 185 | 52

27. Secondary Outcome: Number of Participants With Withdrawal Bleeding From Cycle 1 to Cycle 13
Description: Withdrawal bleedings were defined as bleedings while a participant takes placebo tablets.
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 343
participants
  Cycle 1 | 274
  Cycle 2 | 314
  Cycle 3 | 307
  Cycle 4 | 295
  Cycle 5 | 289
  Cycle 6 | 285
  Cycle 7 | 229
  Cycle 8 | 259
  Cycle 9 | 245
  Cycle 10 | 250
  Cycle 11 | 246
  Cycle 12 | 243
  Cycle 13 | 241

28. Secondary Outcome: Percentage of Participants With Non-heavy Intracyclic Bleeding From Cycle 1 to Cycle 6
Description: Non-heavy bleeding was defined as those other than heavy bleeding (i.e. spotting, light, or normal bleeding).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 349 | 65
Percentage of participants
  Cycle 1 | 90.3 | 89.5
  Cycle 2 | 97.4 | 100.0
  Cycle 3 | 91.1 | 100.0
  Cycle 4 | 87.9 | 100.0
  Cycle 5 | 87.8 | 80.0
  Cycle 6 | 92.5 | 100.0

29. Secondary Outcome: Percentage of Participants With Non-heavy Intracyclic Bleeding From Cycle 1 to Cycle 13
Description: Non-heavy bleeding was defined as those other than heavy bleeding (i.e. spotting, light, or normal bleeding).
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 349
Percentage of participants
  Cycle 1 | 90.3
  Cycle 2 | 97.4
  Cycle 3 | 91.1
  Cycle 4 | 87.9
  Cycle 5 | 87.8
  Cycle 6 | 92.5
  Cycle 7 | 90.4
  Cycle 8 | 100.0
  Cycle 9 | 87.5
  Cycle 10 | 100.0
  Cycle 11 | 100.0
  Cycle 12 | 100.0
  Cycle 13 | 90.3

30. Secondary Outcome: Percentage of Participants With Non-heavy Withdrawal Bleeding From Cycle 1 to Cycle 6
Description: Non-heavy bleeding was defined as those other than heavy bleeding (i.e. spotting, light, or normal bleeding).
Time Frame: Up to Cycle 6 (168 days) with 28 days per cycle
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 349 | 65
Percentage of participants
  Cycle 1 | 90.1 | 87.0
  Cycle 2 | 90.8 | 94.7
  Cycle 3 | 91.2 | 87.9
  Cycle 4 | 92.2 | 92.6
  Cycle 5 | 92.7 | 88.9
  Cycle 6 | 90.9 | 88.5

31. Secondary Outcome: Percentage of Participants With Non-heavy Withdrawal Bleeding From Cycle 1 to Cycle 13
Description: Non-heavy bleeding was defined as those other than heavy bleeding (i.e. spotting, light, or normal bleeding).
Time Frame: Up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 349
Percentage of participants
  Cycle 1 | 90.1
  Cycle 2 | 90.8
  Cycle 3 | 91.2
  Cycle 4 | 92.2
  Cycle 5 | 92.7
  Cycle 6 | 90.9
  Cycle 7 | 91.3
  Cycle 8 | 91.1
  Cycle 9 | 91.0
  Cycle 10 | 90.8
  Cycle 11 | 91.9
  Cycle 12 | 93.8
  Cycle 13 | 93.8

32. Secondary Outcome: Change in Serum Carbohydrate Antigen-125 (CA-125) From Baseline to Cycle 6
Description: CA125 is a laboratory parameter giving an indication of having tumor, whose elevated levels that were defined by a lab suggest a potential tumor.
Time Frame: From baseline up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS(Participants with data at Cycle 6)
Measure: Mean (Full Range); unit: Units/mL
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 281 | 56
Units/mL | -4.33 [-134.8 to 46.1] | -5.50 [-102.6 to 3.2]

33. Secondary Outcome: Change in Serum CA-125 From Baseline to Cycle 13
Description: as for outcome 32
Time Frame: From baseline up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Mean (Full Range); unit: Units/mL
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 254
Units/mL | -4.66 [-135.5 to 90.0]

34. Secondary Outcome: Change in Serum C-reactive Protein (CRP) From Baseline to Cycle 6
Description: CRP is a laboratory parameter giving an indication of inflammation, whose elevated level suggests a potential inflammation.
Time Frame: From baseline up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS(Participants with data at Cycle 6)
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 281 | 56
mg/dL | 0.159 [-0.83 to 7.98] | 0.000 [-1.62 to 1.37]

35. Secondary Outcome: Change in Serum CRP From Baseline to Cycle 13
Description: as for outcome 34
Time Frame: From baseline up to Cycle 13 (364 days) with 28 days per cycle
Population: as for outcome 3
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 254
mg/dL | 0.014 [-0.90 to 1.99]

36. Post Hoc Outcome: Change in Total Dysmenorrhea Score at Final Evaluation in Subgroups (1): From Baseline to Cycle 6
Description: as for outcome 4
Time Frame: Baseline and up to Cycle 6 (168 days) with 28 days per cycle
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (6 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Number analyzed (Participants) | 349 | 65
scores on a scale
  age: < 30 years | -2.4 (1.68) | -2.2 (1.64)
  age: >= 30 years | -2.2 (1.52) | -2.1 (1.69)
  weight: < 50 kg | -2.0 (1.58) | -2.3 (1.76)
  weight: >= 50kg | -2.5 (1.61) | -2.0 (1.60)
  functional dysmenorrhea | -2.4 (1.64) | -2.3 (1.54)
  organic dysmenorrhea | -2.0 (1.45) | -1.3 (1.91)
  with medical surgical history | -2.3 (1.61) | -2.0 (1.69)
  without medical surgical history | -2.4 (1.54) | -2.4 (1.60)
  with previous medication | -2.3 (1.61) | -2.1 (1.66)
  with pregnancy history | -2.2 (1.67) | -2.1 (1.68)
  with birth history | -2.0 (1.71) | -2.4 (1.83)
  total dysmenorrhea score at baseline 3/4 | -1.9 (1.37) | -1.9 (1.37)
  total dysmenorrhea score at baseline 5/6 | -3.0 (1.73) | -2.6 (2.04)

37. Post Hoc Outcome: Change in Total Dysmenorrhea Score at Final Evaluation in Subgroups (1): From Baseline to Cycle 13
Description: as for outcome 4
Time Frame: Baseline and up to Cycle 13 (364 days) with 28 days per cycle
Population: FAS (note: no participants were treated with the DRSP 3 mg/EE 30 µg combination beyond 6 cycles)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles)
Number analyzed (Participants) | 349
scores on a scale
  age: < 30 years | -2.5 (1.67)
  age: >= 30 years | -2.4 (1.70)
  weight: < 50 kg | -2.1 (1.68)
  weight: >= 50kg | -2.7 (1.65)
  functional dysmenorrhea | -2.6 (1.70)
  organic dysmenorrhea | -2.1 (1.59)
  with medical surgical history | -2.5 (1.72)
  without medical surgical history | -2.5 (1.64)
  with previous medication | -2.5 (1.69)
  with pregnancy history | -2.1 (1.75)
  with birth history | -1.9 (1.76)
  total dysmenorrhea score at baseline 3/4 | -2.0 (1.48)
  total dysmenorrhea score at baseline 5/6 | -3.2 (1.75)

ADVERSE EVENTS:
Arm/Group | DRSP 3 mg/EE 20 µg (13 Cycles) | DRSP 3 mg/EE 30 µg (6 Cycles)
Serious Adverse Events (participants affected / at risk) | 5/355 | 0/65
Other Adverse Events (participants affected / at risk) | 335/355 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRSP 3 mg/EE 20 µg (13 Cycles) (N=355) | DRSP 3 mg/EE 30 µg (6 Cycles) (N=65)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRSP 3 mg/EE 20 µg (13 Cycles) (N=355) | DRSP 3 mg/EE 30 µg (6 Cycles) (N=65)
Abdominal pain lower (Gastrointestinal disorders) | 53 (68) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 13 (17) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (34) | 2 (2)
Blood triglycerides increased (Investigations) | 29 (33) | 2 (3)
Constipation (Gastrointestinal disorders) | 19 (20) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 24 (35) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 124 (268) | 20 (42)
Headache (Nervous system disorders) | 215 (679) | 39 (81)
Menorrhagia (Reproductive system and breast disorders) | 16 (21) | 4 (7)
Metrorrhagia (Reproductive system and breast disorders) | 97 (235) | 9 (23)
Nasopharyngitis (Infections and infestations) | 182 (339) | 34 (44)
Nausea (Gastrointestinal disorders) | 128 (217) | 25 (37)
Plasminogen increased (Investigations) | 18 (18) | 7 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 3 (3)
Vomiting (Gastrointestinal disorders) | 22 (24) | 4 (4)
Vulvovaginal candidiasis (Infections and infestations) | 19 (20) | 0 (0)
Seasonal allergy (Immune system disorders) | 35 (38) | 4 (4)
Breast discomfort (Reproductive system and breast disorders) | 13 (15) | 5 (5)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 55 (82) | 11 (11)
Protein S decreased (Investigations) | 9 (9) | 6 (6)
Thrombin-antithrombin III complex increased (Investigations) | 35 (39) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 3 (3) | 4 (4)
Genital haemorrhage (Reproductive system and breast disorders) | 97 (194) | 14 (26)
Coagulation test abnormal (Investigations) | 70 (71) | 12 (12)
Procedural pain (Injury, poisoning and procedural complications) | 19 (25) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will confirm the contents before disclosure.